CLINICAL TRIAL: NCT04652973
Title: Evaluation of Atherosclerotic Plaques in Abdominal CT Studies
Status: Active, not recruiting | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10000123; 000123-CC
Record Dates: First submitted 2020-12-03; First posted 2020-12-04 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08-27

CONDITIONS: Prostatic Neoplasms
Keywords: CT measurement; CVD; CT coronary angiogram; clinical biomarkers; Natural History
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1/Prostate cancer dataset: Biopsy-proven prostate cancer patients who have abdomen CT studies that were available in the clinical PACS (picture archiving system) in the Clinical Center.
- 2/Multiphase CT dataset: Men or women of all age and race, who have Multiphase abdomen-pelvic CT studies that were available in the PACS.

SUMMARY:
Background:

Fat and calcium can build up as plaque in artery walls. The Agatston score measures plaque using computed tomography (CT) that does not use an injected contrast agent. Plaque in the arteries of the pelvis and abdomen is linked to cardiovascular disease (CVD) risk factors. It also may affect cancer. But abdominal CTs use a contrast agent (CECT). Therefore, the Agatston score cannot be used. Researchers want to find a way to measure plaque in CECTs. This will help them use abdominal CTs to measure plaque without extra radiation.

Objective:

To measure atherosclerotic plaques on CECT in a group of males.

Eligibility:

Men ages 30-90 with prostate cancer (proven with biopsies) who have abdomen CT studies in the PACS (picture archiving system) in the Clinical Center. Also, men or women of all ages who have multiphase abdomen and pelvic CT studies that are in the PACS.

Design:

This study will use data gathered since 1/1/2013. Data will also be taken from protocol 03-CC-0128 and clinical trials 15-C-0124, 16-C-0048, 14-C-0112, and 04-C-0274. Participants from these studies have allowed their samples to be used in the future.

Participants will be found via keyword searches on NIH databases. Their CT and MRI scans will be used. Data such as age, race, disease, and treatment will be used. Results of other tests may be used.

The plaque in participants abdomen and iliac arteries will be measured. It will be compared with biomarkers related to CVD and prostate cancer, such as weight, age, and race.

This study will take place at one site. Data will be stored on secure computers. Printouts will be kept in locked rooms.

DETAILED DESCRIPTION:
Evaluation of Atherosclerotic Plaques in Prostate Cancer Patients.

Study Description:

This study measures atherosclerotic plaques in the vessels of prostate cancer patients in contrast-enhanced computed tomography (CECT), then finds correlation between the plaque and clinical biomarkers. These biomarkers include laboratory tests, pathologic findings, underlying risk factors, demographic information, and outcomes of the patient.

Objectives:

Primary objective: Measure atherosclerotic plaques on contrast-enhanced computed tomography (CECT).

Secondary objective: Find correlation between plaque measurement and clinical biomarkers of prostate cancer patients.

Study Population:

Up to 1,000 NIH Clinical Center patients.

Description of Sites/Facilities conducting research:

NIH Clinical Center

Study Duration:

10 years

ELIGIBILITY:
* INCLUSION CRITERIA:

The study will use existing radiologic data.

EXCLUSION CRITERIA:

NONE

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two separate study populations were recruited. The "Prostate cancer dataset" consisted of biopsy-proven prostate cancer patients who have abdomen CT studies that were available in the clinical PACS (picture archiving system) in the Clinical Center. Men of all ages and races are included. The "Multiphase CT dataset" consisted of men or women of all age and race, who have Multiphase abdomen-pelvic CT studies that were available in the PACS.
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2030-08-30 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
1/Measure atherosclerotic plaques | End of study
  Measure atherosclerotic plaques on contrast-enhanced computed tomography (CECT)

SECONDARY OUTCOMES:
2/Plaque measurement and clinical biomarkers correlation | End of study
  Find correlation between plaque measurement and clinical biomarkers of prostate cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Summers, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000123-CC.html